CLINICAL TRIAL: NCT05813028
Title: the Effect of the Interactive Nurse Support Program, Developed as a Mobile Application, on Patient Outcomes in Colorectal Cancer Patients Receiving Chemotherapy During the Covid-19 Process
Brief Title: The Effect of a Mobile Application on Patient Outcomes in Colorectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, burcu ağdemir, research assistant, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Burcu24ankara
Record Dates: First submitted 2023-01-17; First posted 2023-04-14 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Nursing
Keywords: mobile application; Colorectal Cancer; nursing; symptom management
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): As an intervention, the mobile application called KRK-İnHED will be installed on the patients' phones. Patients in the experimental group will be interviewed the day before chemotherapy starts.
  Personal Information Form, Multidimensional Perceived Social Support Scale, Quality of Life Scale, Beck Anxiety Scale will be filled in these patients.
  Mobile application will be installed on the patient's phone by the researcher. The patient will be registered to the program by creating a user name.
  The patient will be given 15-20 minutes of online training on the use of the mobile application.
  The mobile application will be applied for a total of 12 weeks for 4 cycles (1 cycle/3 weeks) from the first day of chemotherapy treatment.
  Interventions: Other: a Mobile Application
- control group (No Intervention): Patients in the control group who will not have a mobile application installed on their phones will receive standard care.

INTERVENTIONS:
Other: a Mobile Application — Patients will use the mobile application for 6 weeks after receiving the first course of chemotherapy. The Multidimensional Scale of Perceived Social Support, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module, Beck Anxiety Scale will be administered when they come to the hospital for their 2nd course of chemotherapy. Patients will use the mobile application for 6 more weeks after receiving the second chemotherapy course. 3. The scales will be reapplied when they come to the hospital for a chemotherapy course. Patients will continue to use the mobile application for three more weeks after receiving their 4th and final cure. When the patients come to the outpatient clinic control in the 12th week, the use of the mobile application will be terminated and the Mobile Application Efficiency Evaluation Form will be applied together with the other scales.
  Other Names: KRK-İnHed
  Arms: experimental group

SUMMARY:
The aim of this study is to determine the effect of the interactive nurse support program developed as a mobile application on patient outcomes (symptom management, quality of life, perception of social support and anxiety) in colorectal cancer patients receiving chemotherapy during the COVID-19 process; It was planned in a randomized controlled, single-blind design. In the study, a mobile application will be designed for colorectal cancer patients with the content created in line with the literature. In the application, the "about COVID-19" module, which includes information for colorectal cancer patients during the COVID-19 process, the "learning module" in which the symptoms and suggestions for colorectal cancer patients receiving chemotherapy are included, the "discussion" module where patients can share their knowledge and experiences with each other, The "ask the expert" module, where nurses and physicians can ask questions, will be comprised of the "lived stories" module and the communication sections, which include interview videos made with individuals who are in remission only after completing the treatment related to the disease. A pretest consisting of Personal Information Form, Multidimensional Perceived Social Support Scale EORTC QLQ-C30 and CR29 Quality of Life Scale, ECOG Performance Scale and Beck Anxiety Scale will be administered to all patients included in the study. The mobile application will be installed on the phones of the patients in the experimental group and they will be used for 12 weeks. Patients in the control group will receive standard care during this process and no intervention will be made. In the sixth and twelve weeks, all participants will be given a posttest. The change in symptom management, quality of life, perceived social support and anxiety levels of the experimental group after mobile application use will be evaluated.

DETAILED DESCRIPTION:
Type of Research:

The research was randomized controlled, analytically planned.

Research Hypotheses:

H0-1: The interactive nurse support program developed with the mobile application in colorectal cancer patients receiving chemotherapy during the COVID-19 process has no effect on the quality of life of the patients.

H0-2: The interactive nurse support program developed with the mobile application in colorectal cancer patients receiving chemotherapy during the COVID-19 process has no effect on the social support perceived by the patients.

H0-3: The interactive nurse support program developed with the mobile application in colorectal cancer patients receiving chemotherapy during the COVID-19 process has no effect on the anxiety levels of the patients.

H0-4: The interactive nurse support program developed with a mobile application has no effect on symptom management in colorectal cancer patients receiving chemotherapy during the COVID-19 process.

Population and Sample of the Research:

The population of the research will be the colorectal cancer patients followed in the Ankara City Hospital Medical Oncology Department Outpatient Clinics.

Calculating Sample Size When previous similar studies on sample size were examined, no similar research could be found in terms of sample characteristics and measurement tools. For this reason, after reaching 10 people in the intervention and control groups, the minimum number of people to be included in the sample will be calculated by performing a power analysis from the research results.

In order to determine the sample size, a similar study (Zhu et al. 2018) was examined, but it was seen that the measurement tools were different. For this reason, after reaching 10 people in the research and control group, power analysis will be made with the G. Power program and the minimum number of people to be sampled will be calculated. It is aimed to increase the number of samples in order to increase the power of the research by guaranteeing the minimum number of people that will constitute the sample size.

Randomization Method:

Among the patients who applied to Ankara City Hospital Medical Oncology Department Outpatient Clinics with the diagnosis of colorectal cancer to receive chemotherapy treatment, patients who meet the criteria for inclusion in the study will be determined. In order to prevent possible interaction between patients who meet the inclusion criteria of the study, data wiil be collected from the control group first, according to the order of admission to the hospital, and after the target number is reached, data will be collected from the patients in the intervention group.

Data Collection Forms

1. Personal Information Form
2. Memorial Symptom Assessment Scale (MSDS)
3. EORTC QLQ-C30 and CR29 Quality of Life Scale
4. Multidimensional Scale of Perceived Social Support (MSPSS)
5. ECOG Performance Scale
6. Beck Anxiety Scale
7. Mobile Application Evaluation Form

Pre-Application:

In order to evaluate the intelligibility and usability of the mobile application and data collection forms created for the interactive nurse support program, a preliminary application was made with 5 patients who met the criteria for inclusion in the study among the patients who applied to Ankara City Hospital Medical Oncology Department Outpatient Clinics with the diagnosis of Colorectal Cancer for chemotherapy treatment. will be done. After the preliminary application, necessary changes will be made in the mobile application and data collection forms. Patients included in the pre-application scope will not be included in the study sample.

Application of Research:

Part 1: Development of Mobile Application 1.1.Developing the Content of the Mobile Application The content of the mobile application will be created by the researcher as a result of extensive literature research. The content created will be submitted to expert opinion, including 1 oncologist, 1 surgical oncology specialist, 4 nurse lecturers, 1 psychiatrist, 1 psychologist, 1 Turkish linguist and 2 oncology nurses. At the same time, the content of the mobile application will be examined by 3 colorectal cancer patients and its comprehensibility will be evaluated. As a result of expert opinions and patient evaluations, arrangements will be made in the content of the mobile application and the mobile application will be finalized.

The content of the mobile application will consist of 5 parts:

* COVID 19 Information Module
* Learning Module
* Discussion Module
* Ask the Expert Module
* Lived Stories Module

Part 2: Implementation of Mobile Application and Collection of Data

* Patients with colorectal cancer who apply to the Department of Medical Oncology will be identified.
* Patients with colorectal cancer who meet the inclusion criteria will be determined (ECOG Performance Scale will be applied at this stage).
* At the beginning of the study, patients who are planned to be included in the study will be informed verbally and in writing about the study and it will be ensured that Informed Consent Forms are filled and signed according to their acceptance status.
* The first day of chemotherapy will be determined for patients who meet the criteria for inclusion in the study and accept to participate in the study. An appointment will be made one day before the chemotherapy treatment and data collection forms will be applied (day 0).

Applications for the Patients in the Experimental Group:

* Interviewing the patients in the experimental group the day before the start of chemotherapy (day 0); Personal Information Form, Multidimensional Perceived Social Support Scale, Quality of Life Scale, Beck Anxiety Scale will be filled.
* The mobile application will be installed on the patient's phone by the researcher. The patient will be registered to the program by creating a changeable user name.
* The patient will be given 15-20 minutes of online training on the use of the mobile application.
* The mobile application will be applied for a total of 12 weeks during 4 cycles of chemotherapy (1 cycle/3 weeks) from the first day of chemotherapy treatment.
* The patient will record the symptoms appearing since the first chemotherapy treatment (symptom type, frequency and severity) in the mobile application, and watch the relevant video recording according to the symptom experienced from the symptom management videos. The patient will be informed that he can record more than one symptom and watch all the videos as many times as he wants. Information texts on patient colorectal cancer and coronavirus will also be accessible at any time. This section covers the "Learning Module" of the mobile application.
* In addition to the video recording, which includes the management initiatives related to the symptom experienced by the patient, the patient will convey his/her individual questions to the researcher by text message or phone call, according to his/her preference. According to the method of conveying the patient's question, the patient's question will be answered by the researcher with the same method. As soon as written messages are sent, they will appear on the researcher's phone screen and the patient will be answered within 1 hour at the latest. If necessary according to the content of the questions regarding the treatment, care or symptom management submitted by the patient, the questions will be directed by the researcher to the oncology physician, who is the other manager in the Ask the Specialist module. The response from the physician will be communicated to the patient. This section covers the "Ask an Expert Module" of the mobile application.
* A reminder message will be sent to the patients who do not register their symptoms and log in to the system during the day, as of 20:00.
* Patients will be able to enter the Discussion Module according to their preferences and share their experiences and opinions with other patients in the control group who had the same experiences. This section covers the "Discussion Module" of the mobile application.
* Patients will be able to watch video recordings containing interviews with patients who have had the same experience and have come to the end of their treatment, whenever they want and as many times as they want. This section covers the "Lived Stories Module" of the mobile application.
* Patients will use the mobile application for 6 weeks after receiving the first course of chemotherapy. The Multidimensional Scale of Perceived Social Support, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module, Beck Anxiety Scale will be administered when they come to the hospital for the 2nd course of chemotherapy (week 6). Patients will use the mobile application for 6 more weeks after receiving the second chemotherapy course. Within these 6 weeks, they will have received the 2nd course of chemotherapy in the 3rd week. 3. The Multidimensional Scale of Perceived Social Support, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module, Beck Anxiety Scale will be re-administered when they come to the hospital for a course of chemotherapy (Week 6). In the second 6 weeks (week 9), patients will have received their 4th chemotherapy course. Patients will continue to use the mobile application for three more weeks after receiving their 4th and final cure. When the patients come to the outpatient clinic at the 12th week, the use of the mobile application will be terminated and the Multidimensional Scale of Perceived Social Support, Memorial Symptom Rating Scale, EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module, Beck Anxiety Scale and Mobile Application Effectiveness Evaluation Form (Appendix 8) will be applied.

Applications for the Patients in the Control Group:

* Patients in the control group who will not have mobile applications installed on their phones will receive standard care.
* The following forms will be filled in by interviewing the patients in the control group the day before chemotherapy starts (day 0).
* Personal Information Form
* Multidimensional Scale of Perceived Social Support
* EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module
* Beck Anxiety Scale
* When the patients come to the outpatient clinic to receive their 3rd course of chemotherapy (week 6), the Memorial Symptom Assessment Scale, Social Support Scale, Quality of Life Scale and Anxiety Scale will be administered to the patients.
* When the patients come to the outpatient clinic (week 12), the Memorial Symptom Rating Scale, Social Support Scale, EORTC QLQ-C30 Quality of Life Scale and QLQ-CR29 Module and Anxiety Scale will be re-administered to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Be over 18 years old
* Being diagnosed with stage 0.1,2 colorectal cancer
* Ability to understand and speak Turkish
* ECOG performance score of 0.1 or 2
* Being literate
* Having a mobile phone with an Android processor and being able to use it effectively
* First time receiving chemotherapy

Exclusion Criteria:

* Presence of a diagnosed psychiatric illness
* Having received previous chemotherapy
* Diagnosis of metastatic colorectal cancer
* ECOG performance score of 3 and 4
* Simultaneous radiation therapy with chemotherapy
* Visual, auditory, mental or neurological disability
* Taking part in another research that will affect the research results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Change of EORTC QLQ-C30 Quality of Life Scale and QLQ- CR29 Module score at baseline and one week later fisrt,second,third and forth chemothraphy. | the first measure will be made before chemotherapy. The second, third,forth and fifth measurement will be madeone week after the first second, third and forth chemotherapy. respectively
  EORTC QLQ-C30 Version 3.0 Quality of Life Scale is a scale developed by EORTC and used in cancer patients. Content validity and reliability study was conducted in Turkey by Beşer and Öz, Cronbach's alpha coefficient was r= 0.9014. The first 28 of the 30 items in the scale are of four-point Likert type and the items are evaluated as Never: 1, A little bit: 2, Quitely: 3, A lot: 4 points. In the 29th question of the scale, the patient is asked to evaluate his health on a scale of 1 to 7 (1: very poor and 7: excellent), and in the 30th question, the patient's overall quality of life is asked. High functional scale and general health status scale scores of the patients; A low symptom scale score indicates a high quality of life. EORTC QLQ CR 29 is an adapted quality of life scale for colorectal cancer. All 29 items in the scale are in four-point Likert type and the items are evaluated as Never: 1, A little: 2, Quitely: 3, A lot: 4 points.
Change of memorial symptom assesment Scale score at baseline and one week later fisrt,second,third and forth chemothraphy. | the first measure will be made before chemotherapy. The second, third,forth and fifth measurement will be madeone week after the first second, third and forth chemotherapy. respectively
  The Memorial Symptom Assessment Scale was developed by Portenoy et al. (1994). The validity and reliability of the scale were made by Yıldırım et al. (2011), and the Cronbach α coefficient was found to be 0.84. The scale has 32 items and allows to evaluate the frequency and severity of the symptoms experienced by cancer patients. While the 'frequency' and 'severity' levels of the symptoms are answered as a 4-point likert, the 'distress' levels are answered as a 5-point likert. The MSAS total score is obtained by averaging the 32 symptom scores. Each symptom score is calculated by averaging the frequency, severity, and degree of distress. Higher values indicate higher frequency, severity, and distress.
Change of Multidimensional Scale of Perceived Social Support Scale score at baseline and one week later fisrt,second,third and forth chemothraphy. | the first measure will be made before chemotherapy. The second, third,forth and fifth measurement will be madeone week after the first second, third and forth chemotherapy. respectively
  The Multidimensional Scale of Perceived Social Support was developed by Zimet et al. (Zimet et al. 1988) and the Turkish validity and reliability of MSPSQ was performed by Eker et al. (Eker et al., 1995). The Multidimensional Scale of Perceived Social Support subjectively evaluates the adequacy of social support from three different sources. This scale is a scale consisting of 12 items. It includes 3 groups related to the source of the support, each of which consists of 4 items. These; family, friends and a special person. Each item was rated using a 7-point scale. In the group treated as a special person; Persons such as dating, relatives, neighbors, doctors and nurses are included. The Turkish reliability of the scale was found to be 0.88 Cronbach'sα coefficient. Any score between 12 and 84 can be obtained from the scale, and a high score indicates a high perceived social support.
Change of Beck Anxiety Inventory score at baseline and one week later fisrt,second,third and forth chemothraphy. | the first measure will be made before chemotherapy. The second, third,forth and fifth measurement will be madeone week after the first second, third and forth chemotherapy. respectively
  Beck Anxiety Inventory is a 21-item self-assessment scale developed by Aeron T. Beck in 1988. Ulusoy et al. It was translated into Turkish and validated in 1998 by The items in the scale describe the subjective, somatic and panic symptoms of anxiety. All item scores are summed as "0=none, 1=mild, 2=moderate, 3=severe" for each item. The scale is evaluated over a total of 63 points, and a high score indicates a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: doğan uncu, professor, Study Director — ankara bilkent central hospital
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No